CLINICAL TRIAL: NCT01154920
Title: Randomized Phase II Trial Contrasting Weekly Paclitaxel, Carboplatin and Cetuximab (PCC) With Cetuximab, Docetaxel, Cisplatin and Fluorouracil (C-TPF) in Previously Untreated Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Paclitaxel, Carboplatin and Cetuximab (PCC) With Cetuximab, Docetaxel, Cisplatin and Fluorouracil (C-TPF) in Previously Untreated Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0885; NCI-2012-01773 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and Neck Cancer; HNSCC; Paclitaxel; Carboplatin; Cetuximab; Docetaxel; Taxotere; Cisplatin; Platinol-AQ; Platinol; CDDP; Fluorouracil; 5-FU; Adrucil; Efudex; chemotherapy; radiation; Chemoradiotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Paclitaxel; Carboplatin; Cetuximab; Docetaxel; Cisplatin; Fluorouracil; Radiotherapy; Drug Therapy; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PCC Group + RT (Experimental): Group A: Paclitaxel, Carboplatin and Cetuximab (PCC) Induction + Radiation (RT)
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Cetuximab; Radiation: Radiotherapy (RT)
- PCC Group + RT + Chemotherapy (Experimental): Group A: Paclitaxel, Carboplatin and Cetuximab (PCC) Induction + Radiation (RT) + Chemotherapy
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Cetuximab; Radiation: Radiotherapy (RT); Other: Chemotherapy
- C-TPF Group + RT (Experimental): Group B: Cetuximab, Docetaxel, Cisplatin and Fluorouracil (C-TPF) Induction + Radiation (RT)
  Interventions: Drug: Cetuximab; Drug: Docetaxel; Drug: Cisplatin; Drug: Fluorouracil; Radiation: Radiotherapy (RT)
- C-TPF Group + RT + Chemotherapy (Experimental): Group B: Cetuximab, Docetaxel, Cisplatin and Fluorouracil (C-TPF) Induction + Radiation (RT) + Chemotherapy
  Interventions: Drug: Cetuximab; Drug: Docetaxel; Drug: Cisplatin; Drug: Fluorouracil; Radiation: Radiotherapy (RT); Other: Chemotherapy

INTERVENTIONS:
Drug: Paclitaxel — 135 mg/m^2 weekly, Weeks 1 - 6
  Other Names: Taxol
  Arms: PCC Group + RT; PCC Group + RT + Chemotherapy
Drug: Carboplatin — AUC of 2 weekly, Weeks 1 - 6
  Other Names: Paraplatin
  Arms: PCC Group + RT; PCC Group + RT + Chemotherapy
Drug: Cetuximab — PCC Arm: 400 mg/m^2 by vein over about 1-2 hours on Day 1; 250 mg/m^2 weeks 2 - 6.
  C-TPF Arm: 250 mg/m2 weeks 2, 4, 5, 7 and 8.
  Other Names: Erbitux; C225; IMC-C225
Drug: Docetaxel — 75 mg/m^2 by vein over 1 hour on Day 1 of each 21 day cycle for 3 cycles of induction therapy
  Other Names: Taxotere
  Arms: C-TPF Group + RT; C-TPF Group + RT + Chemotherapy
Drug: Cisplatin — 100 mg/m^2 by vein over 1-3 hours on Day 1 of each 21 day cycle for 3 cycles of induction therapy
  Other Names: Platinol-AQ; Platinol; CDDP
  Arms: C-TPF Group + RT; C-TPF Group + RT + Chemotherapy
Drug: Fluorouracil — 700 mg/m^2 continuous infusion Days 1-4 on Day 1 of each 21 day cycle for 3 cycles of induction therapy
  Other Names: 5-Fluorouracil; 5-FU; Adrucil; Efudex
  Arms: C-TPF Group + RT; C-TPF Group + RT + Chemotherapy
Radiation: Radiotherapy (RT) — Radiation about 2-4 weeks after induction therapy, Monday through Friday for about 7 weeks, or as recommended by the treating radiologist.
  Other Names: Radiation Therapy; RT
Other: Chemotherapy — PCC group receives 6 and C-TPF group receives 3 chemotherapy treatment cycles. If receiving radiation + chemotherapy, weekly Cisplatin 40 mg/m^2 by vein over 1-3 hours or Carboplatin AUC 2 by vein over 1 hour beginning 2 to 3 weeks after conclusion of induction program.
  Other Names: Chemoradiotherapy
  Arms: C-TPF Group + RT + Chemotherapy; PCC Group + RT + Chemotherapy

SUMMARY:
The goal of this clinical research study is to learn which chemotherapy combination is more effective in treating locally advanced head and neck squamous cell carcinoma. The side effects of these combinations will also be studied.

DETAILED DESCRIPTION:
Treatment on this study consists of 2 parts. The first part of your treatment is called induction chemotherapy and will last for 6-9 weeks, depending on which group you are in. The second part of treatment will be radiation therapy (either with or without chemotherapy). The type of treatment you will receive depends on the site and stage of the disease.

Study Drugs:

Paclitaxel, carboplatin, and 5-fluorouracil are designed to block cancer cells from dividing, which may cause them to die.

Docetaxel is designed to stop the growth of cancer cells, which may cause the cells to die. It may also damage blood vessels in tumor tissue.

Cisplatin has a platinum atom at its center. The platinum is supposed to poison the cancer cells, which may cause them to die.

Cetuximab is designed to prevent or slow down the growth of cancer cells by blocking proteins inside the cancer cell, called the epidermal growth factor receptor (EGFR).

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. There is an equal chance of being assigned to either group.

* If you are in Group A, you will receive cetuximab, paclitaxel, and carboplatin.
* If you are in Group B, you will receive cetuximab, docetaxel, cisplatin, and 5-fluorouracil.

Part 1 Study Drug Administration:

Group A:

During induction, you will receive cetuximab, paclitaxel, and carboplatin by vein once a week for 6 weeks. During Week 1, the cetuximab infusion will last about 2 hours. During Weeks 2-6, the cetuximab infusion will last about 1 hour. Following the cetuximab infusion, you will receive paclitaxel over about 1 hour followed by carboplatin over about 1 hour.

Your vital signs will be monitored before, during, and after the cetuximab infusion.

Group B:

During induction, you will receive cetuximab, docetaxel, and cisplatin by vein. You will also receive 5-fluorouracil as a non-stop infusion over 4 days through an infusion pump. This pump is portable so that you can have this treatment on an outpatient basis.

On Day 1 of each 21-day cycle:

* You will receive cetuximab over about 1-2 hours.
* You will receive docetaxel over about 1 hour.
* You will receive cisplatin over about 1-3 hours
* You will then begin receiving 5-fluorouracil. This infusion will be non-stop over the next 4 days.

On Day 2 of each cycle, you will receive saline (salt water) to prevent dehydration.

On Days 5-10 of each cycle, you will take antibiotics, by mouth, to prevent infection. Your doctor will tell you what type of antibiotic to take.

On Day 8 of each cycle, you will receive cetuximab over about 1 hour.

You will have 3 cycles of induction therapy.

Other drugs may be given before you receive the study drugs to prevent side effects. You will be closely monitored for side effects during the infusions in the clinic setting before you will be allowed to leave.

Part 1 Study Visits:

Every week:

* You will have a physical exam, including measurement of your weight.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* You will be asked about any drugs you may be taking.
* You will be asked about any side effects you may be having.

After you have completed your induction therapy, you will have a CT scan, MRI scan, and/or a PET-CT to check the status of the disease.

Part 2 Study Drug Administration:

Before you begin radiation, you will have a dental exam.

You will begin either radiation with chemotherapy or radiation without chemotherapy. Your doctor will decide which treatment is best for you.

All participants will begin radiation about 2-4 weeks after induction therapy. You will receive radiation Monday through Friday for about 7 weeks, or as recommended by the treating radiologist.

If you are receiving radiation with chemotherapy, you will receive carboplatin or cisplatin every week while you are receiving radiation. If you receive cisplatin, it will be given by vein over about 1-3 hours. If you are given carboplatin, it will be given by vein over about 1 hour.

Part 2 Study Visits:

Every week:

* You will have a physical exam.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* Your skin and the lining of your mouth will be checked for sores.

Follow-Up Phase:

About 6 weeks after you finish all treatments:

* You will have a physical exam.
* You will have a chest x-ray.
* You will be asked about any side effects you may be having.
* You will be asked about any drugs you are taking.
* Your skin and the lining of your mouth will be checked for sores.

If you were in Group B, you will have a CT scan, MRI scan, and/or PET/CT scan at 6 weeks (+/- 14 days) after you have completed radiation/chemoradiation to check the status of the disease.

If you were in Group A, you will have a CT scan, MRI scan, and/or PET/CT scan at 9 weeks (+/- 14 days) after you have completed radiation/chemoradiation to check the status of the disease.

Six (6), 12, and 24 months after you finish treatment, you will have a videofluoroscopic to check your swallowing. You will complete a separate consent form for this procedure. You will also complete the questionnaire about your day-to-day activities.

All participants will have clinic visits every 3 months for 2 years. At these visits:

* You will have a physical exam.
* You will have a chest x-ray.
* You will be asked about any side effects you may be having.
* You will be asked about any drugs you are taking.
* If your doctor thinks it is needed, you will have additional tests/procedures performed.

After the Year 2, follow up will be done per standard of care. You will be contacted by a member of the study team by phone or by letter and asked about you how you are doing and if you have received any other treatment for cancer.

Length of Study:

You will remain on treatment for about 15-16 weeks. If, during that time, the disease gets worse or you experience intolerable side effects, you will be taken off study.

This is an investigational study. All of the study drugs are FDA approved and commercially available. The combination of these drugs when given to patients with locally advanced head and neck squamous cell carcinoma is investigational.

Up to 128 patients will take part in this multicenter study. Up to 100 will be enrolled MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with biopsy-proven squamous cell carcinoma of the oropharynx, oral cavity, nasopharynx, hypopharynx, or larynx.
2. Biopsy material sufficient for HPV status determination available
3. Patients should have stage IV disease, stage T0-4 N2b-2c/3 M0 (for nasopharynx patients, stage N1 is eligible). Measurable disease in either the T or N site by RECIST is required.
4. Patients with stage Tx primary disease are eligible if there is N2b-c/3 lymphadenopathy
5. ECOG PS 0-1
6. Age >/= 18 years
7. Patients should have adequate bone marrow function defined as an absolute peripheral granulocyte count (AGC >/= 1500 cells/mm^3 and platelet count >/= 100,000 cells/mm^3; adequate hepatic function with bilirubin </= ULN (excluding Gilbert's disease), AST and ALT may be up to 2.5 x ULN if alkaline phosphatase is normal. Alkaline phosphatase may be up to 4 x ULN if AST and ALT are normal. In determining eligibility the more abnormal of the two values (AST or ALT) should be used.
8. Creatinine clearance >/=40 ml/min determined by 24 hour collection or nomogram:CrCl male = (140 - age) x (wt in kg)/serum Cr x 72 or CrCl female = 0.85 x (CrCl male)
9. Patients should have no serious acute or chronic co-morbid condition, or acute infection, which in the judgment of the attending physician would affect administration of the induction chemotherapy regimens.
10. Patients must sign a study-specific informed consent form

Exclusion Criteria:

1. Histology other than squamous cell carcinoma
2. Proven distant metastases (below the clavicle) by clinical or radiographic measures
3. ECOG>1
4. Prior chemotherapy, within the previous 3 years
5. Prior radiotherapy to the head and neck
6. Prior cetuximab therapy or prior therapy with any other drug that targets the EGFR pathway
7. Initial surgical resection rendering the patient clinically and radiologically disease free
8. Simultaneous primary invasive cancers, excluding superficial non-melanoma skin cancers
9. Patients with a history of another malignancy (excluding non melanoma skin cancers, and cancers treated > 3 years prior for which patient remains continuously disease free
10. Men and women of childbearing potential (WOCBP) unwilling to consent to using effective contraception while on treatment and for at least 3 months thereafter
11. Women who are pregnant or breastfeeding
12. Pre-existing peripheral neuropathy CTCAE Grade 2 or worse
13. Hemoglobin < 8.0g/dL
14. Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2010-07-09 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Progression-Free Survival (PFS) | 2 Years
  PFS defined as the time from the first day of treatment until the date of objective progressive disease (PD) (locoregional or distant) or death (by any cause in the absence of PD is first reported.

CONTACTS AND LOCATIONS:
Overall Officials: Renata Ferrarotto, MD, Study Chair — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org